CLINICAL TRIAL: NCT05216276
Title: Robotic Versus Conventional Minimal-invasive Inguinal Hernia Repair - a Prospective, Randomized and Blinded Clinical Trial
Brief Title: Robotic vs. Conventional Minimal-invasive Inguinal Hernia Repair
Acronym: ROGER-RCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Clarunis - Universitäres Bauchzentrum Basel (Other); St. Claraspital AG (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-01655
Record Dates: First submitted 2021-12-30; First posted 2022-01-31 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Hernia, Inguinal; Robotic Surgical Procedures
MeSH Terms: conditions — Hernia, Inguinal | interventions — tetraethylpyrazine

STUDY DESIGN:
Intervention Model Description: Patients with indication for inguinal hernia repair are randomized to get a robotic TAPP (rTAPP) or a conventional TEP. Results will be compared primarily pain after 24h hours.
Who Masked: Participant, Outcomes Assessor
Masking Description: patient and assessor blinded study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEP (Active Comparator): Patient with uni- or bilateral inguinal hernia receiving a laparoscopic totally extra-peritoneal (TEP) inguinal hernia repair.
  Interventions: Procedure: TEP
- rTAPP (Experimental): Patient with uni- or bilateral inguinal hernia receiving a robotic transabdominal preperitoneal (TAPP) inguinal hernia repair.
  Interventions: Procedure: rTAPP

INTERVENTIONS:
Procedure: TEP — Laparoscopic totally extra-peritoneal (TEP) inguinal hernia repair
  Arms: TEP
Procedure: rTAPP — robotic transabdominal preperitoneal (TAPP) inguinal hernia repair
  Arms: rTAPP

SUMMARY:
Minimal invasive techniques have become a well established approach for inguinal hernia repair over the last decade in developed countries. Different techniques such as total extraperitoneal endoscopic hernioplasty (TEP) and transabdominal preperitoneal hernia repair (TAPP) have been described. These studies show comparable results in short and long term outcome. Robotic inguinal hernia surgery enables an even more precise dissection within the preperitoneal layer thus preserving the nerves of the lateral abdominal wall. This may translate into a reduced level of acute and chronic postoperative pain as previously reported by retrospective case series. The role of robotic surgery for inguinal hernia repair in regard of postoperative pain and recovery has not been investigated in randomized and blinded clinical studies yet. With this randomized and blinded trial the investigators compare robotic TAPP (rTAPP) to conventional TEP with a decreased pain level shortly after surgery as primary outcome (numeric rating scale - NRS). A reduced postoperative NRS for pain may translate into faster recovery and less chronic pain, secondary endpoints include comparison of pain in a longer course (short-form inguinal pain questionnaire (sf-IPQ)), quality of life / health status (Baseline Short Form-12 (SF-12), Carolinas Comfort Scale (CCS)), complications (Comprehensive Complication Index - CCI), rate of recurrence, , economic impact in terms of costs of surgery per patient, for the institution, the sick leave and the cost-effectiveness of health intervention (SF-6D, EQ-5D, ICECAP-O). Also included are ergonomics for the surgeon (NASA TLX).

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age and able to understand and give their informed consent for the study.
* Primary unilateral or bilateral hernia

Exclusion Criteria:

* Recurrent hernia
* with previous open abdominal surgery at or below the umbilicus
* need of an open inguinal hernia repair (patient's preference, unable to undergo general anesthesia, unable to tolerate pneumoperitoneum)
* liver disease defined by the presence of ascites
* end-stage renal disease requiring dialysis
* unable to give informed consent
* need of an emergency surgery
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain 24 hours post surgery measured on a numeric rating scale (NRS 0-10) | 24 hours
  Pain at coughing 24 hours after surgery measured on a numeric rating scale (NRS 0-10) while coughing

SECONDARY OUTCOMES:
Pain 2 hours post surgery measured on a numeric rating scale (NRS 0-10) | 2 hours
  NRS 2 hours post surgery
Pain 7 days post surgery measured on a numeric rating scale (NRS 0-10) | 7 days
  NRS 7 days post surgery
Pain 30 days post surgery measured on a numeric rating scale (NRS 0-10) | 30 days
  NRS 30 days post surgery
EQ-5D-5L (European Quality of Life - 5 Dimension - 5 Level) questionnaire | 24hours, 7 and 30 days, 6 and 12 months
  EQ-5D-5L 24hours, 7 and 30 days, 6 and 12 months; minimum score = 5, max = 25, lower is better
SF-6D (Short Form - Dimension) questionnaire | 24hours, 7 and 30 days, 6 and 12 months
  SF-6D 24hours, 7 and 30 days, 6 and 12 months; minimum score = 0.0, max = 1.0, higher is better
ICECAP-O (ICEpop CAPability measure for Older people) questionnaire | 24hours, 7 and 30 days, 6 and 12 months
  ICECAP-O 24hours, 7 and 30 days, 6 and 12 months; minimum score = 5, max = 20, higher is better
Intraoperative complications | During surgery
Name and Dosage of pain medication intraoperativ | During surgery
  Amount of intraoperative pain medication
Procedure time | During surgery
  Procedure time
Time in the OR block | During surgery
  Time in the OR block
Time measured in hours patients are in the outpatient clinic until discharge | 24 hours
  For day surgery hours in outpatient clinic until discharge
Time measured in days patients are hospitalized after surgery | 7 days
  For hospitalized patients postoperative stay in days
Pain medication postoperative | 12 months
  Prescribed and actually taken pain medication postoperative 24 hours, 7 days and 30 days, 6 and 12 months after surgery
Postoperative morbidity | 30 days
  Postoperative morbidity classified according to the Dindo-Clavien classification and scored according to the Comprehensive complication index (CCI) up to 30 days after surgery
Recurrence rate | 12 months
  Recurrence rate 6 and 12 months postoperative
SF-12 (Short Form) | 12 months
  SF-12 30 days, 6 months, and 12 months postoperative; The SF-12 Health Survey is a 12-item patient completed questionnaire to measure general health and well-being. It includes a physical and mental status component score; each ranging from 0-100. Low values represent a poor health state and high values represent a good health state.
Carolinas Comfort Scale (CCS) | 12 months
  Carolinas Comfort Scale (CCS) 30 days, 6 months, and 12 months postoperative; minimum score = 8, max = 48, higher is better
Ergonomics for the surgeon | 1 day
  Ergonomics for the surgeon measured by NASA TLX
Costs per patients | 30 days
  Costs for surgery per patient according to the accounting department
Sick leave | 12 months
  ays until resumption of work or days until resumption of activities of daily life, and estimated sick leave by patient
Costs for sick leave | 12 months
  Costs for sick leave (days multiplied by average daily costs of sick leave in Switzerland according to the Swiss National Accident Insurance Fund (SUVA))
Type of labor including the relative activity level | 1 day
  Type of labor including the relative activity level (sedentary work, light work, medium work, heavy work, very heavy work, retired/unemployed) according to US Code of Federal Regulations § 404.1567 Physical exertion requirement

CONTACTS AND LOCATIONS:
Overall Officials: Fiorenzo V Angehrn, Dr. med., Principal Investigator — Clarunis AG
Locations (1):
- Clarunis AG, Basel, Basel-Landschaft, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Angehrn FV, Susstrunk J, Schneider R, Baltzer K, Muller BP, Baur J, Steinemann DC. Robotic versus laparoscopic minimally invasive inguinal hernia repair: randomized clinical trial (the ROGER trial). Br J Surg. 2025 Dec 24;113(1):znaf283. doi: 10.1093/bjs/znaf283. PMID 41511872
- [Derived] Angehrn FV, Neuschutz KJ, Baur J, Schneider R, Wilhelm A, Stoll L, Susstrunk J, von Flue M, Bolli M, Steinemann DC. Robotic Versus Conventional Minimal-Invasive Inguinal Hernia Repair: Study Protocol for a Prospective, Randomized and Blinded Clinical Trial. Int J Surg Protoc. 2022 Jun 6;26(1):27-34. doi: 10.29337/ijsp.175. eCollection 2022. PMID 35794884